CLINICAL TRIAL: NCT03574168
Title: Phase I Study of the Safety and Efficacy of CD19-CAR-T Cells in Patients With Relapsed or Refractory Acute B-cell Lymphoblastic Leukemia (R/R B-ALL)
Brief Title: CD19-CAR-T Cells in Patients With R/R B-ALL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioceltech Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-ALL-001-v2; ChiCTR1800016541 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2018-06-11; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-CAR-T Cells (Experimental): Subjects will receive CD19-CAR-T Cells on Day 0 : 100% of total dose.
  Interventions: Biological: CD19-CAR-T Cells

INTERVENTIONS:
Biological: CD19-CAR-T Cells — T cells purified from the PBMC of subjects or subjects' relatives which depends on their conditions, transduced with 4-1BB/CD3-ζ lentiviral vector, expanded in vitro for future administration.

SUMMARY:
This is a single center, single arm, open-lable phase 1 study to determine the safety and efficacy of autologous or donor-derived allogeneic T cells expressing CD19 chimeric antigen receptors (referred to as "CD19-CAR-T cells") in patients with relapsed or refractory acute B-cell lymphoblastic leukemia (R/R B-ALL).

DETAILED DESCRIPTION:
Primary objective:

To investigate the safety and efficacy of autologous or HLA-haploidentical Allo-CD19-CAR-T cells in the treatment of patients with relapsed or refractory acute B-cell lymphoblastic leukemia.

Secondary objective:

To Assess the patient's quality of life after receiving the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain Informed Consent Form (ICF) voluntarily signed by the patient;
2. Age 3-70 years old;
3. Primary resistant or relapsed B-cell line acute lymphoblastic leukemia;
4. B cells are positive for CD19 expression;
5. Peripheral blood tumor cell load <50%; 6. KPS score >50 points;

7. Normal liver and kidney function; 8. Normal heart function; 9. Good follow-up compliance; 10. Women of childbearing age (15-49 years old) must have a pregnancy test within 7 days before treatment and have a negative result; Men and women with fertility should agree to use effective contraception to ensure that during the study period and following 3 months after treatment the women will not get pregnant.

Exclusion Criteria:

1. Patients with non-B cell acute leukemia;
2. Organ failure: Heart: Grade III and IV Liver: Class C with Child-Turcotte liver function classification Kidney: Renal failure and uremia Lung: severe respiratory failure Brain: Disabilities
3. Active infection;
4. Human immunodeficiency virus (HIV) positive;
5. Acute and chronic graft-versus-host disease (GVHD)> Level 1；
6. Pregnant or lactating women;
7. Patients do not agree to use effective contraception during the treatment period and following 3 months;
8. Patients who participated in other clinical studies at the same time;
9. The researcher believes that there are other factors that are not suitable for inclusion in or influence the subject's participation in or completion of the study;
10. Long-term use greater doses of hormones than physiological doses.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-20 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | Up to Day90 after the CD19-CAR-T cell infusion
  The percentage of participants who achieved complete remission (CR) over all participants (CRR).
  The percentage of participants who achieved partial remission (PR) over all participants (PRR).

SECONDARY OUTCOMES:
The amount of CAR-T cells remaining in vivo | 2 years after cell infusion.
  Measure and analyze monthly
The lifetime of CAR-T cells remaining in vivo | 2 years after cell infusion.
  Measure and analyze monthly

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, MD, PhD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided